CLINICAL TRIAL: NCT00059267
Title: Prevention of Recurrent Hepatitis B After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: NIH HBV-OLT (completed); U01DK057577 (NIH)
Record Dates: First submitted 2003-04-22; First posted 2003-04-23 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B; Cirrhosis; Acute Liver Failure; Hepatocellular Carcinoma
MeSH Terms: conditions — Hepatitis B; Fibrosis; Liver Failure, Acute; Carcinoma, Hepatocellular | interventions — hepatitis B hyperimmune globulin; Lamivudine; adefovir dipivoxil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: HBIG, Epivir, Hepsera

SUMMARY:
Hepatitis B accounts for approximately 5000 deaths per year in the United States. Liver transplantation offers the only hope for patients who develop end-stage liver disease. Early results of liver transplantation for hepatitis B were poor with recurrence rate of 80% and 1-year survival of only 50%. Recent studies found that preventive therapy using hepatitis B immune globulin (HBIG) or antiviral medications such as lamivudine can reduce the recurrence rate to roughly 30% with accompanying improvement in survival. However, HBIG when given as intravenous infusion in high doses is very expensive, while long-term use of lamivudine is associated with drug resistance. Some studies found that preventive therapy using both HBIG and lamivudine may decrease recurrence rate to less than 10% but the dose and duration of HBIG needed when used in combination with lamivudine is not clear. Adefovir, a new antiviral medication, is effective against lamivudine resistant hepatitis B but its role in liver transplantation is uncertain because of the risk of kidney damage. Many studies showed that the risk of recurrent hepatitis B is related to the viral load before transplant. Thus, it may be possible to tailor the preventive therapy according to the risk. The aim of this study is to establish the most cost-effective preventive therapy for recurrent hepatitis B after liver transplantation.

ELIGIBILITY:
Inclusion criteria: adult patients listed for liver or liver-kidney transplant for hepatitis B.

Exclusion criteria: patients with contraindications to use of prophylactic antiviral therapy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients listed for liver or combined liver-kidney transplantation for hepatitis B including hepatitis B cirrhosis, hepatitis B liver cancer and fulminant hepatitis B.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2001-03 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Lok, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Degertekin B, Han SH, Keeffe EB, Schiff ER, Luketic VA, Brown RS Jr, Emre S, Soldevila-Pico C, Reddy KR, Ishitani MB, Tran TT, Pruett TL, Lok AS; NIH HBV-OLT Study Group. Impact of virologic breakthrough and HBIG regimen on hepatitis B recurrence after liver transplantation. Am J Transplant. 2010 Aug;10(8):1823-33. doi: 10.1111/j.1600-6143.2010.03046.x. Epub 2010 Mar 23. PMID 20346062